CLINICAL TRIAL: NCT06906341
Title: An Open-label, Global, Multi-Arm Study to Evaluate the Efficacy and Safety of Relacorilant in Combination With Different Treatment Regimens in Patients With Gynecological Cancers (BELLA)
Brief Title: Relacorilant in Combination With Different Treatment Regimens in Patients With Gynecological Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORT125134-557
Record Dates: First submitted 2025-04-01; First posted 2025-04-02 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Neoplasms; Endometrial Cancer
Keywords: Genital Neoplasms, Female; Neoplasms by Site; Fallopian Tube Diseases; Ovarian Diseases; Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Peritoneal Neoplasms; Paclitaxel; Albumin-Bound Paclitaxel; Ovarian; Peritoneal or Advanced Fallopian Tube Cancer; High Grade; Platinum Resistant; Relacorilant; Bella; Nab-paclitaxel; Bevacizumab; Endometrial Neoplasm; Endometrial
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms; Endometrial Neoplasms; Genital Neoplasms, Female; Neoplasms by Site; Fallopian Tube Diseases; Ovarian Diseases; Neoplasms | interventions — relacorilant; 130-nm albumin-bound paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A: Relacorilant in Combination with Nab-paclitaxel and Bevacizumab (Experimental): In Arm A, patients with platinum-resistant ovarian cancer will receive the combination of relacorilant with nab-paclitaxel and bevacizumab.
  Interventions: Drug: Relacorilant 150 mg once daily (QD); Drug: Nab-paclitaxel 80 mg/m^2; Drug: Bevacizumab 10 mg/kg
- Arm B: Relacorilant in Combination with Nab-Paclitaxel and Bevacizumab (Experimental): In Arm B, patients with platinum-sensitive ovarian cancer who have progressed while receiving treatment with a polymerase inhibitor will receive relacorilant in combination with nab-paclitaxel and bevacizumab.
  Interventions: Drug: Relacorilant 150 mg once daily (QD); Drug: Nab-paclitaxel 80 mg/m^2; Drug: Bevacizumab 10 mg/kg
- Arm C: Relacorilant in Combination with Nab-Paclitaxel (Experimental): In Arm C, patients with previously-treated advanced, recurrent, or metastatic endometrial cancer will receive relacorilant in combination with nab-paclitaxel.
  Interventions: Drug: Relacorilant 150 mg once daily (QD); Drug: Nab-paclitaxel 80 mg/m^2

INTERVENTIONS:
Drug: Relacorilant 150 mg once daily (QD) — Relacorilant is administered under fed conditions as capsules for oral dosing on the day before, the day of, and the day after nab-paclitaxel infusion.
  Other Names: CORT125134
Drug: Nab-paclitaxel 80 mg/m^2 — Nab-paclitaxel is administered as IV infusion on Days 1, 8, and 15 of each 28-day cycle.
Drug: Bevacizumab 10 mg/kg — Bevacizumab is administered as IV infusion on Days 1 and 15.
  Arms: Arm A: Relacorilant in Combination with Nab-paclitaxel and Bevacizumab; Arm B: Relacorilant in Combination with Nab-Paclitaxel and Bevacizumab

SUMMARY:
This is a Phase 2, open-label, global, multi-arm study to evaluate efficacy and safety of relacorilant in combination with other treatments in patients with gynecological cancers.

DETAILED DESCRIPTION:
This study is designed with the goal to add additional arms as new treatments become available. All arms will follow an independent and parallel design.

For Arms A and B, study treatment will comprise relacorilant combined with nab-paclitaxel, and bevacizumab and will begin on Cycle 1 Day 1 (C1D1). Each patient will receive relacorilant 150 mg administered orally under fed conditions, once daily for 3 consecutive days on the day before, the day of, and the day after nab-paclitaxel infusion (in Cycle 1 relacorilant is only given on 2 consecutive days, starting on C1D1), in combination with nab-paclitaxel (80 mg/m^2 intravenously [IV]) administered on Days 1, 8, and 15 of each 28-day cycle. Bevacizumab (10 mg/kg IV once every 2 weeks [Q2W]) will be administered on Days 1 and 15 of each 28-day cycle. Study treatment for Arm C will be similar to Arm A but does not include bevacizumab. Patients will receive treatment until they reach a protocol-defined event of progressive disease (PD), experience an unmanageable toxicity, or until other treatment discontinuation criteria are met.

ELIGIBILITY:
Inclusion Criteria:

Arms A and B

* Histologic diagnosis of epithelial ovarian, primary peritoneal, or fallopian-tube carcinoma
* Arm A Only: Platinum-resistant disease
* Arm B Only: Platinum-sensitive disease who had progression while receiving treatment with a poly(ADP-ribose) polymerase (PARP) inhibitor
* Life expectancy of ≥3 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Able to swallow and retain oral medication
* 1 to 3 lines of prior systemic anticancer therapy
* Adequate organ function
* Negative pregnancy test for patients of childbearing potential

Arm C

* Stage III or IV, recurrent, or metastatic endometrial cancer
* Life expectancy of ≥3 months
* ECOG performance status of 0 or 1
* Able to swallow and retain oral medication
* Prior treatment with a platinum agent and an approved anti-Programmed Cell Death Ligand 1 (PD[L]1) antibody
* 1 to 2 lines of prior systemic anticancer therapy for endometrial cancer
* Must consent to provide an available formalin-fixed paraffin-embedded (FFPE) tumor tissue block or recently cut sections
* Adequate organ function
* Negative pregnancy test for patients of childbearing potential

Exclusion Criteria:

Arm A and B

* Arm A Only: Has progressed while receiving weekly paclitaxel or nab-paclitaxel
* Prior enrollment in a clinical trial of relacorilant
* Prior anticancer therapy related toxicities not resolved to grade ≤1
* Any surgery within 4 weeks prior to enrollment
* Wide-field radiation to more than 25% of marrow-bearing areas
* Medical conditions requiring chronic or frequent treatment with corticosteroids
* Concurrent treatment with mifepristone or other glucocorticoid receptor modulators
* Peripheral neuropathy from any cause >Grade 1
* Hypertension: ≥150 mm Hg systolic or ≥100 mm Hg diastolic
* Uncontrolled condition(s) which, may confound the results of the trial or interfere with the patient's safety or participation
* Bowel obstruction ≤12 weeks prior to study entry
* Ascites or pleural effusions requiring therapeutic paracentesis
* Untreated or symptomatic central nervous system metastases
* History of other malignancy within 3 years prior to enrollment
* Has received a live vaccine within 30 days prior to the study start date

Arm C

* Has progressed while receiving weekly paclitaxel or nab-paclitaxel
* Prior enrollment in a clinical trial of relacorilant
* Prior anticancer therapy related toxicities not resolved to grade ≤1
* Any surgery within 4 weeks prior to enrollment
* Wide-field radiation to more than 25% of marrow-bearing areas
* Medical conditions requiring chronic or frequent treatment with corticosteroids
* Concurrent treatment with mifepristone or other glucocorticoid receptor modulators
* Peripheral neuropathy from any cause >Grade 1
* Uncontrolled condition(s) which, may confound the results of the trial or interfere with the patient's safety or participation
* Bowel obstruction ≤12 weeks prior to study entry
* Ascites or pleural effusions requiring therapeutic paracentesis
* History of other malignancy within 3 years prior to enrollment
* Has received a live vaccine within 30 days prior to the study start date
* Patients with central nervous system metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Date of first dose until PD or death, up to 18 months
  To evaluate PFS as the time from enrollment until first documented progressive disease (PD) by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as determined by the Investigator, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Date of first dose until PD or death, up to 18 months
  To evaluate the proportion of patients with measurable disease at Baseline who attain complete response (CR) or partial response (PR) by RECIST version 1.1.
Best Overall Response Rate (BOR) | Date of first dose until PD or death, up to 18 months
  To evaluate the BOR by RECIST version 1.1 recorded from the date of enrollment until PD or death
Duration of Response (DOR) | Time of first objective response until PD or death, up to 18 months
  To evaluate DOR as the time from the first CR or PR to first objectively documented PD or death, whichever comes first.
Clinical Benefit Rate (CBR) | Week 24
  To evaluate CBR as the proportion of patients who attain CR, PR, or stable disease (SD) at Week 24 as per RECIST version 1.1.
Overall Survival (OS) | Date of first dose up to 6, 12, and 18 months
  To evaluate the probability of OS survival at 6, 12, and 18 months.
Number of patients with one or more adverse events | Date of first dose up to 30 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Pai, MD, MS, Study Director — Corcept Therapeutics
Locations (45):
- United States (14):
  - 150, Palo Alto, California
  - 014, San Francisco, California
  - 544, Fort Myers, Florida
  - 543, West Palm Beach, Florida
  - 518, Minneapolis, Minnesota
  - 334, Kansas City, Missouri
  - 521, St Louis, Missouri
  - 292, Albuquerque, New Mexico
  - 304, Centerville, Ohio
  - 517, Eugene, Oregon
  - 127, Pittsburgh, Pennsylvania
  - 522, Fairfax, Virginia
  - 300, Norfolk, Virginia
  - 121, Milwaukee, Wisconsin
- Belgium (4):
  - 328, Aalst
  - 326, Charleroi
  - 325, Hasselt
  - 108, Leuven
- France (6):
  - 306, Lille
  - 307, Nancy
  - 310, Nice
  - 324, Pierre-Bénite
  - 323, Plérin
  - 308, Toulouse
- Germany (3):
  - 519, Aachen
  - 255, Berlin
  - 520, Kempten
- Italy (7):
  - 321, Catania
  - 122, Milan
  - 516, Milan
  - 295, Pavia
  - 124, Rome
  - 293, Torino
  - 319, Treviso
- Poland (2):
  - 341, Gdynia
  - 329, Siedlce
- South Korea (6):
  - 396, Seoul, Gangnam-gu
  - 397, Gyeonggi-do, Goyang-si
  - 399, Seoul, Jongno-gu
  - 523, Seoul, Seocho-gu
  - 398, Seoul, Seodaemun-gu
  - 403, Seoul, Songpa-gu
- Spain (3):
  - 349, Badalona
  - 115, Barcelona
  - 330, Valencia

IPD SHARING:
Plan to Share IPD: No